CLINICAL TRIAL: NCT06737926
Title: Effects of Sensorimotor Training on Pain Intensity, Perceived Balance Confidence and Functional Exercise Capacity With Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Effects of Sensorimotor Training With Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0204
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy; Breast Cancer Patients
Keywords: Breast Cancer; Chemotherapy-Induced Peripheral Neuropathy; Postural Balance; Sensorimotor Neuropathy; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Experimental Group receiving Sensorimotor Training Exercise. (Experimental): Participants will undergo sensorimotor training exercises targeting balance, pain reduction, and functional exercise capacity.
  Interventions: Behavioral: Sensorimotor Training Exercise
- Group B: Control Group receiving Conventional Exercise Therapy. (Active Comparator): Participants will receive conventional exercise therapy as per standard guidelines.
  Interventions: Behavioral: Conventional Exercise Therapy

INTERVENTIONS:
Behavioral: Sensorimotor Training Exercise — Participants will perform sensorimotor training exercises designed to improve balance, reduce pain intensity, and enhance functional exercise capacity. The program will include progressive exercises focusing on proprioception, neuromuscular coordination, and functional mobility. Sessions will be conducted thrice weekly over 12 weeks, supervised by a physiotherapist.
  Arms: Group A: Experimental Group receiving Sensorimotor Training Exercise.
Behavioral: Conventional Exercise Therapy — Participants will undergo conventional exercise therapy, including stretching, strengthening, and aerobic exercises, based on standard physiotherapy protocols. The therapy aims to maintain joint mobility, reduce stiffness, and improve general physical fitness. Sessions will be conducted thrice weekly over 12 weeks, supervised by a physiotherapist.
  Arms: Group B: Control Group receiving Conventional Exercise Therapy.

SUMMARY:
Chemotherapy-Induced Peripheral Neuropathy (CIPN) is a prevalent and clinically relevant side effect of chemotherapy in breast cancer patients. It occurs in 30-70% of cases. It can cause various sensory and motor symptoms. Specific exercise interventions have proven promising to target relevant symptoms. Therefore, the objective of this study is to determine the effects of Sensorimotor training on pain intensity, perceived balance confidence, and functional exercise capacity with chemotherapy-induced peripheral neuropathy in breast cancer patients.

DETAILED DESCRIPTION:
The study incorporated a single blinded randomized controlled trial conducted at Mayo Hospital, Lahore. It involved 22 participants (N=22) recruited by using non-probability convenience sampling technique according to inclusion criteria and randomly allocated into either of two groups (Experimental group or Control group) using randomizer.org. The participants in experimental group performed sensorimotor training based on progressively challenging balance exercises on unstable surfaces. Participants performed three sets of exercises per session twice a week for 6 weeks, 45 minutes per session. The control group performed conventional exercises such as range of motion, stretching, strengthening, deep breathing and aerobic exercises for 2 times a week for 6 weeks, 45 minutes per session. Pre and post assessment of participants was done on numeric pain rating scale for pain intensity, TUG test for balance, activities-specific balance confidence scale for perceived balance confidence, 6-minute walk test for functional exercise capacity and EORTC QLQ C-30 for quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Females with invasive ductal carcinoma, stages I-III
* Age ranged between 30-65 years
* 3-6 months post breast cancer diagnosis
* Those who have completed chemotherapy treatment and are medically stable
* CIPN symptoms as subjectively assessed by FACT/GOG-Ntx. Score ranges from 0-44 (5). 0 - 10: Minimal or no neurotoxicity symptoms, 11 - 20: Mild neurotoxicity symptoms, 21 - 30: Moderate neurotoxicity symptoms, 31 - 40: Severe neurotoxicity symptoms, 41 - 44: Very severe neurotoxicity symptoms
* For balance testing Fullerton Advanced Balance (FAB) scale was used. 0-19 = high risk of falls, 20-29 = moderate balance impairment, 30-40 = good balance. The cut off value is ≤ 25/40 Points.
* Objective neurological testing such as Achilles and patellar tendon reflexes (1 = agile, 2 = weak, 3 = missing), peripheral deep sensitivity (0=no sensitivity to 8=highest sensitivity), light touch perception (symmetrical or impaired), sense of position (1 = position recognized, 2 = only position of knee recognized, and 3 = no recognition) and lower leg strength (0 = no activity to 5 = normal force) rated on a Likert-scale

Exclusion Criteria:

* Women with additional types of cancer besides breast cancer
* Chronic medical conditions such as poorly controlled diabetes (6)
* Significant neurological (multiple sclerosis) or cardiopulmonary disease (myocardial infarction < 3 months) that may affect performance (6)
* Unstable bone metastasis

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  It is a uni-dimensional subjective measure of pain intensity in adults, including those with cancer pain. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible.
TUG Test | 6 weeks
  It is used to determine the fall risk and measure the progress of balance. Mobility and balance is assessed based on time to complete the test: < 10 seconds = normal. < 20 seconds = good mobility < 30 seconds = walking and balance problems
Activities-Specific Balance Confidence Scale | 6 weeks
  The ABC-Scale is a self-reported assessment of the participant's level of confidence in static and dynamic balance while doing functional activities
6-Minute Walk Test | 6 weeks
  The 6-minute walk test (6MWT) is a standardized field test used to predict cardio-respiratory fitness in healthy individuals, as well as to assess functional exercise capacity and responsiveness to rehabilitation treatments in a variety of patient groups

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) Subscale | 6 weeks
  The FACT/GOG Ntx subscale is designed to measure chemotherapy-induced PN. It contains 11 items covering sensory neuropathy, motor neuropathy, hearing neuropathy, and dysfunction associated with neuropathy
EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) | 6 weeks
  The EORTC QLQ-C30 is composed of nine multi-item scales: 5 functioning scales (physical, role, cognitive, emotional and social), a global QOL scale, and 3 symptom scales (fatigue, pain and nausea/vomiting).
Fullerton Advanced Balance Scale (FAB Scale) | 6 weeks
  It is a screening tool which can be used in different group. It has long form (consisting of 10 tasks) and a short form (consisting of 4 tasks). The scale consists of a 5-point Likert scale from 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, M.phil, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Mayo Hospital Lahore, Lahore, Punjab Province
  - Mayo Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Twice-weekly neuromuscular stimulation training reduced the incidence of chemotherapy-induced peripheral neuropathy compared with standard care, especially among patients taking vinca alkaloids. — https://www.jwatch.org/na57738/2024/08/05/does-neuromuscular-training-help-prevent-chemotherapy